CLINICAL TRIAL: NCT00212511
Title: Prospective Evaluation of Patients With Idiopathic Pulmonary Fibrosis Through an IPF Registry
Brief Title: Evaluation of Patients With Idiopathic Pulmonary Fibrosis (IPF) Through an IPF Registry
Status: Withdrawn | Type: Observational
Why Stopped: Pending more information from PI
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 10386-02 A
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to create a database of demographics and samples in idiopathic pulmonary fibrosis.

ELIGIBILITY:
Inclusion Criteria

1. Male or Female greater or equal to age 18.
2. Referral by physician with the diagnosis of IPF, or interstitial lung disease (IPF considered likely).

Exclusion Criteria

(a) Unwilling or unable to give written informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with interstitial lung disease.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2004-11; Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Determine cellular and molecular determinants of IPF | Long-Term
  An IPF Registry is being established to assemble sufficient patients with IPF (especially in its earliest stage) for phase I therapeutic protocols. The Registry will incorporate demographic and clinical data for natural history studies; second, research data on physiology, high-resolution CT scan, questionnaires, and blood samples for blood banking to be collected every 6 months for prospective studies on pathophysiology; and third, response to standard therapies will be monitored to determine cellular and molecular relationships to clinical outcome and predictors of survival. This is done in order to better determine cellular and molecular determinants of IPF. This cohort will be large enough to commence a separate phase I protocol with molecular strategies of intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Rany Condos, MD, Principal Investigator — NYU School of Medicine, Division of Pulmonary and Critical Care Medicine
Locations (1):
- NYU School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Data has not been analyzed yet.